CLINICAL TRIAL: NCT05992012
Title: Myocardial Infarction Triggers and Onset in Jordan Study (MINTOR) 2
Brief Title: Myocardial Infarction Triggers and Onset in Jordan Study 2
Acronym: MINTOR 2
Status: Terminated | Type: Observational
Why Stopped: Protocol not adopted by study teams
Sponsor: Jordan Collaborating Cardiology Group (Other)
Responsible Party: Sponsor
Other Study IDs: CVAG.MINTOR2.7AUG23
Record Dates: First submitted 2023-08-07; First posted 2023-08-15 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-08

CONDITIONS: Triggers of Acute Myocardial Infarction; Time of Onset of Acute Myocardial Infarction; Long-term Prognosis After Acute Myocardial Infarction
Keywords: Acute myocardial infarction; Acute ST-segment elevation myocardial infarction; Triggers of acute myocardial infarction; Middle East; Prognosis
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A previous study (MINTOR 1) found that 43% of ST elevation myocardial infarction (STEMI) patients in Jordan had a triggering events. Fifteen years later, with changing demographics and in the post covid-19 time, we believe that triggered acute myocardial infarction might have changed in incidence and nature of the triggering events.

DETAILED DESCRIPTION:
The onset of acute ST elevation myocardial infarction (STEMI) is a complex interplay of internal circadian factors and external physical and emotional triggers. These interactions may lead to rupture of an often nonocclusive vulnerable atherosclerotic coronary plaque with subsequent formation of an occlusive thrombus. The onset of MI has a distinct pattern, with peak incidence within the first few hours after awakening, on certain days of the week, and in the winter months. Physical and emotional stresses are important triggers of acute cardiovascular events including MI. Triggering events, internal changes, and external factors vary among different geographical, environmental, and ethnic regions. Life-style changes, pharmacotherapy, and psychologic interventions may potentially modify the response to, and protect against the effects of triggering events.

MINTOR 1 showed that 43% of 900+ Jordanians with STEMI were exposed to a physical or emotional triggers before the onset of the heart attack. It was also found that Friday was the day of the week that witnessed more MIs that other days of the week and that 55% of MIs occurred in the early morning hours.

It is largely unknown if the frequency and types of triggers, onset time of MI, day with peak of MI incidence have changed over time in Jordan with changing population demographics, especially in the post Covid-19 times. These patients will be followed up for 3 years for occurring of incident vascular events.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and above.
* Documented acute ST elevation myocardial infarction.
* Willing to sign an informed consent.
* Available contact numbers for a 3-year follow up

Exclusion Criteria:

* Unwilling to sign an informed consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adults aged 18 years and above admitted with a diagnosis of acute ST elevation myocardial infarction will be asked about the potential presence of a triggering event prior to the heart attack as well the exact timing (hour of the day and the day of the week) when the pain of the heart attack started.
  Furthermore these patients will be followed up for 3 years to study the occurrence of future cardiovascular event at 3 years. These events include all-cause death, myocardial infarction, stroke, heart failure and repeat coronary revascularization (percutaneous of surgical).
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2023-12-24 (Actual); Study Completion 2023-12-25 (Actual)

PRIMARY OUTCOMES:
Triggers of acute myocardial infarction | From date of study enrollment until the date of a documented exposure to a trigger, up to the time of discharge from the hospital (2-5 days).
  Exposure to emotional of physical triggering events before the occurrence of the heart attack
Time of onset of acute myocardial infarction | From date of study enrollment until the date of documenting the day and hour of onset of the heart attach, up to the time of discharge from the hospital (2-5 days)
  Documenting the time of onset of the chest pain that marks the onset of the myocardial infarction (expressed as day of the week (MONDAY to SUNDAY) and time of the day (00:00 hr to 24:00 hr).
Acute cardiovascular events | From date of study enrollment until the date of occurrence of the first cardiovascular event (described above) up to three years after study enrollment.
  Occurrence of death from any cause, myocardial infarction, stroke, heart failure, repeat coronary revascularization (percutaneous or surgical).

CONTACTS AND LOCATIONS:
Overall Officials: Daria Jaara, MD, Study Director — Istishari Hospital
Locations (1):
- Istishari Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Yes
Will send e mails to other tertiary care institutions inviting them to participate in the study
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Immediately after the date of securing an NCT unique number, up to 6 months after that date.